CLINICAL TRIAL: NCT02751749
Title: Chronic Pain and Emotional Problems: a Single Case Study of an Internet Based Self-help Treatment Based on CBT Principles and the Unified Protocol for Transdiagnostic Treatments
Brief Title: A Transdiagnostic Treatment for Comorbid Chronic Pain and Emotional Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Örebro County Council (Other Government); Uppsala County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Matilda Wurm, PhD fellow, Örebro University, Sweden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STARK
Record Dates: First submitted 2016-04-11; First posted 2016-04-26 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Pain and Comorbid Emotional Problems
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Unified Protocol (Experimental): CBT based Internet delivered treatment targeting transdiagnostic vulnerability and maintaining factors for chronic pain and emotional problems.
  Since this is a new target Group, a replicated single case design was used and participants are their own Control Group (no other treatment arms).
  Interventions: Behavioral: Unified Protocol

INTERVENTIONS:
Behavioral: Unified Protocol

SUMMARY:
The study uses a replicated randomized single case design. Participants were 12 individuals with chronic pain problems and residual problems after undergoing a multimodal pain rehabilitation. They also had comorbid emotional problems. Treatment consisted of 10 weeks of Internet delivered, therapist guided CBT based self-help treatment based on the Unified Protocol.

DETAILED DESCRIPTION:
The study uses a replicated randomized single case design. Twelve participants were recruited from three pain clinics and five primary care centers in different municipalities in central Sweden. The clinics and care centers provided addresses and sent a total of 600 letters with information regarding the study to patients who had completed a multimodal pain rehabilitation (MMR) at their facility within the last three years. Participants were also recruited via the Internet through an advertisement on Google Ads that was visible for two months. No reward was offered for taking part in the study. Potential participants were screened and provided demographic information on a secure internet based platform. Afterwards all screened individuals received a telephone call. Excluded individuals were informed about the reason for exclusion and given recommendations regarding alternative treatment options when indicated. Eligible participants were screened further using selected parts of the Mini International Neuropsychiatric Interview. They were also given more information about the study and invited to ask questions. Individuals who met selection criteria were randomized in blocks of four using randomizer.org and half participated in an initial pilot study while half participated in the treatment study reported here. Participants for the treatment study were thereafter randomized to either a short (five week) or a long (10 week) baseline as well as separately randomized to one of five therapists. Therapists were two clinical psychology students in their last year of training, one graduated clinical psychologist, one postgraduate clinical psychology fellow and one certified clinical psychologist. Participants gave written informed consent by sending in a form included in the initial information letter.

Participants were 12 individuals with chronic pain problems. The sample consisted of 9 females (75 %) and 3 males (25 %). Participants' age ranged from 30 to 60 (M= 47, sd= 9). See table 1 for further description of the participants. All participants had completed MMR within the past three years.

Participants for the treatment study filled in baseline measurements at between 3 and 10 time points. Baseline measurements were separated by at least five days. In connection with the last baseline measurement, participants filled out pretreatment measurements and started treatment, consisting of 10 weekly modules. Process measurements were filled out once every module, as well as longer measurements at mid- and post treatment. A follow-up was done via the platform after 3 months. Treatment consisted of 10 weeks of internet delivered, therapist guided CBT based self-help treatment based on the Unified Protocol.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain problems (duration > 3 months)
* Depressive symptoms and/or anxiety symptoms (> 15 points on the Swedish Montgomery Åsberg Depression Schedule (MDRS-S) and/or > 7 points on the Overall Anxiety Symptoms and Impairment Scale, (OASIS))
* MMR within the last three years
* > 18 years
* Fluent in reading and writing Swedish, and
* Internet access.

Exclusion Criteria:

* Ongoing or planned psychological treatment delivered by a psychologist or a psychotherapist
* Planned surgery
* Suicidality
* Severe depression
* Ongoing alcohol or substance abuse, and
* Ongoing psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Overall Depression Severity and Impairment Scale (ODSIS) | an average of 30 weeks
  measures general depression
Overall Anxiety Severity and Impairment Scale (OASIS) | an average of 30 weeks
  measures general anxiety
The question: How intense has your pain been during the last week? | an average of 30 weeks
  one item asking for pain during last week (1-10)

SECONDARY OUTCOMES:
Mini International Neuropsychiatric Interview, MINI | an average of 30 weeks
  diagnostic interview

CONTACTS AND LOCATIONS:
Overall Officials: Matilda Wurm, Principal Investigator — Örebro University, Sweden

IPD SHARING:
Plan to Share IPD: Undecided